CLINICAL TRIAL: NCT00888368
Title: Accuracy of the Transpatellar Tendon Approach to Knee Arthrocentesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DHMC07-0387
Record Dates: First submitted 2009-04-23; First posted 2009-04-27 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Knee Aspiration

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Transpatellar Approach (Experimental)
  Interventions: Procedure: Transpatellar Approach
- Suprapatellar Approach (Active Comparator)
  Interventions: Procedure: Suprapatellar

INTERVENTIONS:
Procedure: Transpatellar Approach — The transpateller approach for the injection of the dye will be used.
  Arms: Transpatellar Approach
Procedure: Suprapatellar — The suprapatellar approach will be used for the injection of the dye.
  Arms: Suprapatellar Approach

SUMMARY:
The purpose of this study is:

* To determine the accuracy of intraarticular placement with the transpatellar tendon approach as compared to the suprapatellar approach. Patients undergoing knee arthroscopy will be consented for study of the injection of the fluid into the joint prior to portal placement or commencement of knee replacement. Patients will be randomized to receive injections via the transpatellar tendon or superolateral approach. Using injectable contrast and fluoroscopy, the placement of injections into the knee will be evaluated for accuracy. Injection attempts with contrast fluid that uniformly coats the articular surface on sagittal and coronal radiographs will be counted as successful. A concentration of contrast fluid in extraarticular fat will be counted as a failure.

Hypothesis: The rate of accuracy of intraarticular placement of the needle tip via the transpatellar tendon approach to knee aspiration is greater than that of the superolateral approach.

* To determine the distribution of contrast material with the transpatellar tendon and superolateral apporaches. Using a previously described evaluation technique of dividing the knee into seven compartments, sagittal and coronal fluoroscopy images will be evaluated to determine the distribution of contrast fluid.

Hypothesis: Contrast injected into the knee via the trasnpatellar tendon approach will penetrate as many compartments of the knee as contrast injected via the superolateral approach.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective arthroscopic surgery of the knee
* age greater than 18 years old and less than 80 years old
* able to consent to a research study

Exclusion Criteria:

* allergy to contrast dye, iodine or shellfish
* currently pregnant
* acute fracture or dislocation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The development of an easier approach to aspirating the knee may lead to improved accuracy of intraarticular needle placement by less experienced practitioners and more "anatomically difficult" knees. | 1 time (intraop)

CONTACTS AND LOCATIONS:
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States